CLINICAL TRIAL: NCT06903910
Title: Investigating the Cholinergic Contribution to Gait Dysfunction in Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, William Alex Dalrymple, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR230410
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Gait; Cholinergic
MeSH Terms: conditions — Parkinson Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Donepezil (Experimental): Patients with Parkinson's disease and gait dysfunction will be enrolled. We will measure gait metrics and obtain an MRI at baseline, then everyone will begin donepezil (5mg nightly for 4 weeks, followed by 10mg nightly). There will be a telephone check in at week 6, then at week 12 they will return for repeat gait metrics
  Interventions: Drug: Donepezil (Aricept)

INTERVENTIONS:
Drug: Donepezil (Aricept) — Donepezil is a cholinesterase inhibitor tablet taken by mouth once nightly

SUMMARY:
People with Parkinson's disease often experience problems with 'gait' and balance. Gait refers to the way a person moves while walking, such as their speed and length of steps. People with Parkinson's may experience slowness of movement, shuffle their feet, or have periods of 'freezing', during which their feet feel like they are stuck to the floor. Some people may struggle to maintain their balance and fall. These symptoms are frequently disabling and can lead to a worse quality of life. The nervous system is your body's messaging system - it helps different parts of your body communicate with one another. Neurotransmitters are chemicals that deliver those messages from one part of the body to another. The purpose of this study is to determine if the use of ARICEPT (Donepezil hydrochloride) improves gait and balance and its relation to the size of an area of the brain called "Cholinergic Nucleus 4" (Ch4). The study team is also studying how degeneration (breakdown and eventual loss) in Ch4 contributes to problems with gait and balance. One way this may happen is through the loss of a chemical in the brain called acetylcholine. Acetylcholine is a neurotransmitter and its activity is associated with alertness, thinking, and the ability to move. Taking a drug that increases acetylcholine, such as ARICEPT, may improve gait and balance. By better understanding this relationship, we may be able to improve the treatment of gait and balance problems in the future.

DETAILED DESCRIPTION:
Background and Rationale Parkinson's disease (PD) is the most common neurodegenerative movement disorder, affecting approximately 1% of people over the age of 60 years.1 As the population ages, the prevalence of PD is expected to double by 2040.2 PD presents with multiple symptoms, including the triad of bradykinesia, cogwheel rigidity, and resting tremor.3 Impairment of gait and balance is another cardinal feature of the disease, and remains poorly responsive to medical therapies.4 Patients with PD often experience reduced gait speed, reduced stride length, slower turns, freezing of gait, and falls.4,5

Although dopaminergic deficiency is considered responsible for most of the motor symptoms of PD, gait dysfunction often responds poorly to dopaminergic therapies.6-8 Recent work has shown that central cholinergic degeneration also plays a key role in development of gait dysfunction in PD.9,10 Degeneration of these projections, arising from Cholinergic Nucleus 4 (Ch4) within the basal forebrain, has been associated with impairments in gait and balance in PD.11-14 Given this evidence, the cholinergic system thus becomes an attractive therapeutic target for gait dysfunction in PD. In fact, expert opinion called for novel application of imaging methods to investigate the cholinergic contribution to gait in PD.15 We propose the use of a novel tool to detect Ch4 degeneration as a way to improve patient selection and therefore therapeutic targeting in gait dysfunction, which currently remains resistant to treatment, worsens disease morbidity, and contributes to rising care costs.

Innovation Assessment of Ch4 degeneration has previously proven challenging - prior studies have relied on cholinergic positron emission tomography (PET) imaging16,17 or transcranial magnetic stimulation to measure short latency afferent inhibition (SAI).18 Conventional imaging techniques, such as computed tomography (CT) or standard magnetic resonance imaging (MRI), are unable to delineate the borders of Ch4 and other cholinergic nuclei within the basal forebrain.19 PET and SAI have the disadvantage of being expensive, not widely available, and with limited clinical use in Parkinson's disease outside of a research setting.

Recently, a novel method based on MRI techniques has been shown to quantify Ch4 degeneration via calculation of basal forebrain grey matter density (GMD) in a two-part manner. First, whole brain voxel-based morphometry (VBM) of grey matter is measured via MRI.20,21 Then, cholinergic basal forebrain probabilistic masks are applied to the VBM results, which allows quantification of regional GMD in Ch4. These cholinergic basal forebrain probabilistic masks were derived from a 2008 study involving imaging and histopathology of 10 different post-mortem brains: cholinergic nuclei were mapped onto the brain MRI, and these nuclei were then mapped onto a commonly-used Montreal Neurological Institute (MNI) stereotactic brain space. Using data from all 10 post-mortem brains, they were able to create a mask in the MNI space showing the probability that a specific cholinergic nucleus (Ch4) lies in a specific location in the MNI space.22 As this process to determine Ch4 GMD is a deterministic algorithm, inter-rater reliability is not a concern (in other words, it will always give the same output when fed the same input). Likewise, intra-patient reliability of Ch4 GMD is excellent.23 Importantly, this MRI technique has been shown to have adequate sensitivity in prior studies of neurodegeneration.24

Our team has previously published a retrospective study investigating the relationship between Ch4 GMD, as measured via this MRI technique, and gait speed in a cohort of patients with PD undergoing workup for deep brain stimulator placement. In this study, we demonstrated that lower Ch4 GMD was associated with reduced gait speed in patients with PD.25 This retrospective result was the impetus for the current proposed trial.

This current study seeks to prospectively support the relationship between Ch4 GMD and gait dysfunction in patients with PD, as well as to provide some preliminary data to inform a future larger-scale trial investigating the relationship between Ch4 GMD and gait response to cholinesterase inhibitors.

The first aim of this project is to gather prospective supporting evidence of what our group has previously shown via retrospective analysis: that lower Ch4 GMD is associated with more gait dysfunction in patients with PD. Our hypothesis is that lower Ch4 GMD will be associated with slower gait speed. We will also investigate other gait metrics, including self-selected gait speed, Timed Up and Go, Cognitive Timed Up and Go, 4-Stage Balance Test, Modified Clinical Test of Sensory Interaction and Balance, Functional Gait Assessment, fall history, and the Freezing of Gait Questionnaire to prospectively determine their relationships and to better define outcome measures for a hypothetical future trial.

The second aim of this project is to gather preliminary data regarding the use of baseline Ch4 GMD to predict improvement in gait with cholinesterase inhibitors. Our hypothesis is that we can see improvement in gait speed, among other gait metrics, in a subset of patients with PD following 12 weeks of donepezil administration. We believe that baseline Ch4 values can be used to identify that specific subset of patients. While this study will not be powered to truly define that relationship, it will provide the necessary preliminary data for a future investigation designed to do just that.

Study Design This proposed study will be done in two parts. First, we plan to enroll 5 patients with PD who are able to ambulate independently, and MRIs will be obtained for Ch4 GMD quantification. Gait metrics as well as other clinical data will be measured by a physical therapist (co-investigator Diane Huss, DPT) and a movement disorders neurologist (the principal investigator), both of whom will be blinded to Ch4 GMD values. We will then analyze the relationship between Ch4 GMD and gait speed, seeking to support our hypothesis that lower Ch4 GMD will be associated with slower gait speed. We will also investigate the relationship between Ch4 GMD and the other gait metrics measured, with a goal of determining which metrics would be best to measure in a hypothetical future trial.

Second, we plan to give these same 5 patients donepezil for 12 weeks, and measure their gait metrics again at the end of the study. Initial screening tests will include electrocardiogram, serum chemistry, and Montreal Cognitive Assessment (MoCA). We will obtain gait metrics at baseline (for part 1 as described above), and then patients will be given donepezil in an unblinded fashion for 12 weeks (5mg nightly for 4 weeks, then 10mg nightly), after which we will again obtain gait metrics. All gait metrics will be measured in the on dopaminergic state, and all doses of anti-parkinsonian medications will be held constant through the 12 weeks of the study. We expect that some of the patients will show improvement in some of the gait metrics, and we hope to also show that baseline Ch4 GMD could potentially be used as a predictor for gait improvement following cholinesterase inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PD by a neurologist as per UK Brain Bank criteria
2. Age 40 or older
3. Clinical evidence of gait dysfunction, as determined by a movement disorders neurologist.
4. Willingness and ability to comply with scheduled visits and study procedures.
5. Actively treated with a stable dose of levodopa or other anti-parkinsonian medications.
6. Able to ambulate without the use of an assistive device.
7. Serum chemistry from blood obtained at screening will need to be free from evidence of renal injury (elevated creatinine) or other significant metabolic abnormalities at the discretion of the examiner within 28 days of study initiation.
8. Subject agrees not to participate in another study with an investigational drug/treatment during this study and for 3 months following study completion.
9. Female subjects must not be breastfeeding and must have a negative serum pregnancy test at Visit 1. Women of childbearing potential (WOCBP) must use one of the following acceptable birth control methods as specified before enrollment and throughout the trial:

   * Surgical sterilization (bilateral tubal occlusion/ligation) prior to signing the informed consent form (ICF).
   * Intrauterine device in place for at least 3 months before the first dose of study drug and throughout the trial.
   * Barrier method (condom or diaphragm) with spermicide for at least 30 days before the first dose of the study drug and throughout the trial.
   * Surgical sterilization of the male partner (vasectomy at least 6 months before the first dose of study drug).
   * Hormonal contraceptives with a barrier method for at least 3 months before the first dose of the study drug and throughout the trial.

Female subjects are not considered to be of childbearing potential if they meet at least one of the following criteria as documented by the Investigator:

* They have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at minimum one menstrual cycle prior to signing the ICF.
* They are postmenopausal, defined as 1 year since the last menstrual period without an alternative medical cause or have a follicle-stimulating hormone (FSH) level in the menopausal range (defined as >20 miU/mL and <122 miU/mL) in women who are not using hormonal contraception or hormonal replacement therapy and are ≥50 years of age.
* For women ≤50 years old, ≥2 years since her last menstrual period without an alternative.

Exclusion Criteria:

1. Current use of donepezil, rivastigmine, galantamine, or memantine
2. Score of 3 or higher on the Anticholinergic Cognitive Burden Scale
3. Presence of a deep brain stimulator, or implantation of a deep brain stimulator during the study
4. Montreal Cognitive Assessment (MoCA) score less than 21
5. Known allergic reactions to donepezil or piperidine derivatives
6. Use of a different investigational drug/treatment within 3 months before the study
7. Presence of bradycardia for bradycardia (<60bpm) and other significant arrhythmias (not counting simple first-degree heart block), severe COPD, severe asthma, peptic ulcer disease, or other severe, acute medical comorbidities that could affect the outcome of the study, for example acute end-stage CHF or acute pneumonia
8. Inability to obtain a brain MRI (presence of ferromagnetic metal inside the body, severe claustrophobia, etc)
9. Impairment in cognitive or decision-making abilities that would impede the participant's ability to consent for themselves. Of note, physical impairment or disability may still require the use of a legally authorized representative or surrogate, and would not in itself be an exclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between Ch4 GMD and gait speed | Baseline
  We hypothesize that lower baseline Ch4 GMD will be associated with slower baseline gait speed

SECONDARY OUTCOMES:
Relationship between baseline Ch4 GMD and gait response to donepezil | From enrollment to the end of treatment at 12 weeks
  We hypothesize that we will be able to see improvement in gait speed (and potentially other gait metrics) following 12 weeks of donepezil administration, at least in some patients. We believe that baseline Ch4 values can be used to identify that specific subset of patients.

CONTACTS AND LOCATIONS:
Overall Officials: William A Dalrymple, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No